CLINICAL TRIAL: NCT07021872
Title: Reducing Loneliness Among Older Adults Through Enhancing Positive Affect: A Randomized Controlled Trial With Ecological Momentary Assessments
Brief Title: Reducing Loneliness Among Older Adults Through Enhancing Positive Affect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: University of Texas at Austin (Other); City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jiang Da, Associate Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-2024-0179
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Loneliness
Keywords: Loneliness; Older Adults; Positive Affect; Behavioral Activation; Randomized Controlled Trials

STUDY DESIGN:
Intervention Model Description: A three-armed randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Affect (Experimental): Participants in the Positive Affect group will receive the Tele-PA Intervention to test the effects of the intervention in reducing loneliness among older adults.
  Interventions: Behavioral: Tele-Positive Affect Intervention
- Behavioral Activation (Experimental): Participants in the Behavioral Activation group will receive the Tele-BA Intervention to test the effects of the intervention in reducing loneliness among older adults.
  Interventions: Behavioral: Tele-Behavioral Activation Intervention
- Friendly Visit (Active Comparator): Participants in the Friendly Visit group will receive the Tele-FV Intervention as an active control.
  Interventions: Behavioral: Tele-Friendly Visit

INTERVENTIONS:
Behavioral: Tele-Positive Affect Intervention — A 4-week intervention consisting of eight skills aimed at enhancing positive affect, delivered via telephone by trained facilitators. Participants will learn skills such as gratitude, mindfulness, and positive reappraisal, with sessions held twice a week.
  Arms: Positive Affect
Behavioral: Tele-Behavioral Activation Intervention — A 4-week intervention designed to promote engagement in meaningful activities, delivered through telephone by trained facilitators. The intervention will include behavior monitoring, activity planning, and social skills enhancement, with sessions held twice a week.
  Arms: Behavioral Activation
Behavioral: Tele-Friendly Visit — An active control condition consisting of telephone-delivered friendly visits. Participants will engage in social conversation and activities to provide companionship without any specific skills training aimed at reducing loneliness. The intervention will be held within 4-week.
  Arms: Friendly Visit

SUMMARY:
This study aims to evaluate the effectiveness of two psychosocial interventions-Tele-Positive Affect (Tele-PA) and Tele-Behavioral Activation (Tele-BA)-compared to active control (telephone-delivered friendly visit, Tele-FV) in reducing loneliness among older adults in Hong Kong.

DETAILED DESCRIPTION:
Loneliness in older adults represents a critical public health challenge, associated with detrimental outcomes including depression, cardiovascular risks, cognitive decline, and elevated mortality. Despite existing interventions, significant gaps persist: most approaches neglect the affective dimension of loneliness, fail to address the core mechanism of perceived discrepancies between expected and actual social relationships, and inadequately account for age-related shifts in socioemotional goals. This randomized controlled trial addresses these limitations by evaluating two theoretically distinct telephone-delivered psychosocial interventions against an active comparator.

The study employs a three-arm design to compare a 4-week Tele-Positive Affect (Tele-PA) intervention grounded in the broaden-and-build theory of positive emotion, which aims at increasing positive affect through eight evidence-based skills (e.g., gratitude, mindfulness, positive reappraisal), and a Tele-Behavioral Activation (Tele-BA) intervention derived from the behavioral explanations of learning theory, focusing on behavior monitoring and strategies, valued activity scheduling, and social skill enhancement. Both are contrasted with Tele-Friendly Visit (FV)-an active control condition comprising matched-frequency neutral conversations devoid of therapeutic components.

Community-dwelling adults aged ≥65 years in Hong Kong with significant loneliness will be randomized to these arms. Using a three-arm, assessor-blinded randomized clinical trial, outcomes will be measured through retrospective surveys and ecological momentary assessments (EMA) at baseline, immediately post-intervention (Week 2), and at 3- and 6-month follow-ups. Primary analyses will examine: 1) the comparative efficacy of Tele-PA and Tele-BA versus the active control in reducing loneliness; 2) differential effectiveness of Tele-PA versus Tele-BA; 3) the mechanisms underlying the effects of Tele-PA and Tele-BA; and 4) the effects of age on the effectiveness.

This research pioneers the integration of affective science with loneliness intervention design while employing EMA to capture mechanistic dynamics. Findings will advance precision approaches for alleviating loneliness in aging populations through scalable, theory-informed strategies.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* proficiency in Cantonese (over telephone)
* experiencing loneliness (defined as a score of ≥ 6 on the 3-item UCLA Loneliness Scale)

Exclusion Criteria:

* cognitive impairments
* psychiatric disorders, learning disabilities, or active suicidal ideation
* currently participating in other psychotherapy or psychosocial interventions aimed at enhancing well-being

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Loneliness measured by the UCLA Loneliness Scale | Baseline, 3-month, and 6-month
  The UCLA Loneliness Scale is a reliable self-assessment tool designed to evaluate feelings of loneliness. Possible scores range from 1 (never) to 4 (always).
Loneliness measured by De Jong Gierveld Loneliness Scale | Baseline, 3-month, and 6-month
  The De Jong Gierveld Loneliness Scale is a validated, self-reported instrument assessing loneliness. Possible scores range from 1 (yes) to 3 (no).
Real-time Experiences on Ecological Momentary Assessment | Baseline and 2-week
  Ecological Momentary Assessment (EMA) is a research method used to collect data in real-time and in the participants' natural environments. It measures momentary loneliness, momentary actual affect examined by the short version of the AVI scale, current and expected locations (e.g., nature, home, public places), as well as details about their current and expected social interactions, including the type (i.e., alone, with spouse, family members), features (e.g., supportiveness, closeness, pleasantness, meaningfulness), and number (i.e., 0, 1, 2, 3, 4, 5, or more than 5). Participants will also report on their current and expected activities, specifying the type (e.g., physical activity, working, cognitive activities) and characteristics (e.g., pleasantness, meaningfulness) of these activities.

SECONDARY OUTCOMES:
Psychological Well-being on 6-point Psychological Well-being Scale | Baseline, 3-month, and 6-month
  The Psychological Well-being Scale is a validated, self-reported instrument assessing Psychological Well-being. Possible scores range from 1 (strongly disagree) to 6 (strongly agree).
Perceived Stress on 5-point Chinese Version of the Perceived Stress Scale | Baseline, 3-month, and 6-month
  The Chinese version of the Perceived Stress Scale is a validated self-report tool used to measure Perceived Stress levels. Possible scores range from 0 (never) to 4 (very often).
Symptoms of Depression on 4-point Chinese Version of Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3-month, and 6-month
  PHQ-9 is a reliable self-report measure designed to evaluate Symptoms of depression. Possible scores range from 0 (not at all) to 3 (nearly everyday).
Symptoms of Anxiety on 4-point Chinese Version of the Generalized Anxiety Disorder Scale | Baseline, 3-month, and 6-month
  The Chinese version of the Generalized Anxiety Disorder Scale is a validated, self-reported instrument assessing Symptoms of depression. Possible scores range from 0 (not feeling at all) to 3 (most of the time).
Cognitive Functioning on the Hong Kong Version of Montreal Cognitive Assessment | Baseline, 3-month, and 6-month
  The Hong Kong version of the Montreal Cognitive Assessment (MoCA-HK) is a validated tool administered by clinicians to evaluate cognitive functioning, especially in older adults. Possible scores range from 0 to 30, with higher scores indicating better cognitive performance.
Perceived Social Support on 7-point Multidimensional Scale of Perceived Social Support | Baseline, 3-month, and 6-month
  The Multidimensional Scale of Perceived Social Support evaluates the social support derived from three key sources: family, friends, and significant others. Respondents rated each item on a 7-point Likert scale, where 1 represents "very strongly disagree" and 7 indicates "very strongly agree."
Social Network on Lubben Social Network Scale at Month 3 and Month 6 | Baseline, 3-month, and 6-month
  The Lubben Social Network Scale is a validated, self-reported instrument assessing the social networks of participants. This scale comprises six items, with three focused on family connections (family subscale) and three addressing friendships (friend subscale). The overall score ranges from 0 to 30, with each subscale spanning from 0 to 15.

OTHER OUTCOMES:
Affective Experience over the Past Week on 30-item Affect Valuation Index (actual affect) (AVI) | Baseline, 3-month, and 6-month
  The Affect Valuation Index (AVI) is a validated, self-reported instrument assessing affective experiences over the past week. It evaluates both the actual emotions experienced and the ideal emotions valued by the individual. Possible scores for each emotion reflect the frequency of experience, typically ranging from 1 (very slightly or not at all) to 5 (extremely or all the time).
Social Network Characteristics on 10-point Social Network Characteristics Scale | Baseline, 3-month, and 6-month
  The Social Network Characteristics Scale will assess the perceived supportiveness, closeness, pleasantness, and meaningfulness of participants' social partners over the past two weeks. Possible scores range from 1 (not at all) to 10 (extremely high). Additionally, participants will report the number of social partners they have engaged with during this same timeframe.
Meaning of Life on 7-point Meaning in Life Questionnaire (MLQ) | Baseline, 3-month, and 6-month
  The MLQ is a reliable self-assessment tool that evaluates individuals' sense of meaning in life. This instrument comprises two subscales: Presence of Meaning and Search for Meaning, with each subscale containing five items. Each subscale has a minimum score of 5 and a maximum score of 35.
Gratitude on 7-point Gratitude Scale Questionnaire-Six Item Form (GQ-6) | Baseline, 3-month, and 6-month
  The GQ-6 is a validated self-report measure that evaluates inclination to recognize, appreciate, and respond to life events with gratitude. Possible scores range from 1 (strongly disagree) to 7 (strongly agree).
Cognitive Reappraisal on 7-point Emotional Regulation Questionnaire (ERQ) | Baseline, 3-month, and 6-month
  The ERQ is a validated, self-reported instrument assessing emotional regulation strategies, specifically cognitive reappraisal (6 items) and expressive suppression (4 items). Possible scores range from 1 (strongly disagree) to 7 (strongly agree).
Self-Efficacy on 4-point General Self-Efficacy Scale (GSE) | Baseline, 3-month, and 6-month
  The GSE is a validated instrument assessing participants' self-reported levels of self-efficacy. This validated instrument consists of 10 items designed to measure individuals' optimistic beliefs regarding their capacity to manage challenging situations. Participants will evaluate each statement using a 4-point Likert scale, where 1 indicates "not at all true" and 4 represents "exactly true."
Mindfulness on 5-point Five Facet Mindfulness Questionnaire | Baseline, 3-month, and 6-month
  The Five Facet Mindfulness Questionnaire is a validated measure assessing levels of mindfulness. Responses will be scored on a 5-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true).

CONTACTS AND LOCATIONS:
Overall Officials: Da Jiang, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu X, Tam WW, Wong PT, Lam TH, Stewart SM. The Patient Health Questionnaire-9 for measuring depressive symptoms among the general population in Hong Kong. Compr Psychiatry. 2012 Jan;53(1):95-102. doi: 10.1016/j.comppsych.2010.11.002. Epub 2010 Dec 28. PMID 21193179
- [Background] Wong A, Xiong YY, Kwan PW, Chan AY, Lam WW, Wang K, Chu WC, Nyenhuis DL, Nasreddine Z, Wong LK, Mok VC. The validity, reliability and clinical utility of the Hong Kong Montreal Cognitive Assessment (HK-MoCA) in patients with cerebral small vessel disease. Dement Geriatr Cogn Disord. 2009;28(1):81-7. doi: 10.1159/000232589. Epub 2009 Aug 11. PMID 19672065
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Verstaen A, Moskowitz JT, Snowberg KE, Merrilees J, Dowling GA. Life Enhancing Activities for Family Caregivers of people with dementia: protocol for a randomized controlled trial of a positive affect skills intervention. Open Access J Clin Trials. 2018;10:1-12. doi: 10.2147/oajct.s150597. Epub 2018 Feb 7. PMID 33981167
- [Background] Orgeta V, Brede J, Livingston G. Behavioural activation for depression in older people: systematic review and meta-analysis. Br J Psychiatry. 2017 Nov;211(5):274-279. doi: 10.1192/bjp.bp.117.205021. Epub 2017 Oct 5. PMID 28982660
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Moskowitz JT, Hult JR, Duncan LG, Cohn MA, Maurer S, Bussolari C, Acree M. A positive affect intervention for people experiencing health-related stress: development and non-randomized pilot test. J Health Psychol. 2012 Jul;17(5):676-92. doi: 10.1177/1359105311425275. Epub 2011 Oct 21. PMID 22021272
- [Background] Moskowitz JT, Cheung EO, Snowberg KE, Verstaen A, Merrilees J, Salsman JM, Dowling GA. Randomized controlled trial of a facilitated online positive emotion regulation intervention for dementia caregivers. Health Psychol. 2019 May;38(5):391-402. doi: 10.1037/hea0000680. PMID 31045422
- [Background] Moskowitz JT, Carrico AW, Duncan LG, Cohn MA, Cheung EO, Batchelder A, Martinez L, Segawa E, Acree M, Folkman S. Randomized controlled trial of a positive affect intervention for people newly diagnosed with HIV. J Consult Clin Psychol. 2017 May;85(5):409-423. doi: 10.1037/ccp0000188. Epub 2017 Mar 23. PMID 28333512
- [Background] Mccullough ME, Emmons RA, Tsang JA. The grateful disposition: a conceptual and empirical topography. J Pers Soc Psychol. 2002 Jan;82(1):112-27. doi: 10.1037//0022-3514.82.1.112. PMID 11811629
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Lindsay EK, Chin B, Greco CM, Young S, Brown KW, Wright AGC, Smyth JM, Burkett D, Creswell JD. How mindfulness training promotes positive emotions: Dismantling acceptance skills training in two randomized controlled trials. J Pers Soc Psychol. 2018 Dec;115(6):944-973. doi: 10.1037/pspa0000134. PMID 30550321
- [Background] Lindsay EK, Young S, Brown KW, Smyth JM, Creswell JD. Mindfulness training reduces loneliness and increases social contact in a randomized controlled trial. Proc Natl Acad Sci U S A. 2019 Feb 26;116(9):3488-3493. doi: 10.1073/pnas.1813588116. Epub 2019 Feb 11. PMID 30808743
- [Background] Leung GT, de Jong Gierveld J, Lam LC. Validation of the Chinese translation of the 6-item De Jong Gierveld Loneliness Scale in elderly Chinese. Int Psychogeriatr. 2008 Dec;20(6):1262-72. doi: 10.1017/S1041610208007552. Epub 2008 Jul 1. PMID 18590603
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Lay JC, Ho YW, Tse DCK, Tse JTK, Jiang D. Misremembering Solitude: The Role of Personality and Cultural Self-Concepts in Shaping Discrepancies Between Recalled and Concurrent Affect in Solitude. J Pers. 2025 Feb;93(1):174-192. doi: 10.1111/jopy.12971. Epub 2024 Aug 16. PMID 39149879
- [Background] Jiang D, Fung HH, Sims T, Tsai JL, Zhang F. Limited time perspective increases the value of calm. Emotion. 2016 Feb;16(1):52-62. doi: 10.1037/emo0000094. Epub 2015 Jul 27. PMID 26214569
- [Background] Jiang D. Feeling Gratitude Is Associated With Better Well-being Across the Life Span: A Daily Diary Study During the COVID-19 Outbreak. J Gerontol B Psychol Sci Soc Sci. 2022 Apr 1;77(4):e36-e45. doi: 10.1093/geronb/gbaa220. PMID 33284976
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Heinrich LM, Gullone E. The clinical significance of loneliness: a literature review. Clin Psychol Rev. 2006 Oct;26(6):695-718. doi: 10.1016/j.cpr.2006.04.002. Epub 2006 Jun 19. PMID 16952717
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Folkman S. The case for positive emotions in the stress process. Anxiety Stress Coping. 2008 Jan;21(1):3-14. doi: 10.1080/10615800701740457. PMID 18027121
- [Background] Folkman S. Positive psychological states and coping with severe stress. Soc Sci Med. 1997 Oct;45(8):1207-21. doi: 10.1016/s0277-9536(97)00040-3. PMID 9381234
- [Background] Ferster CB. A functional anlysis of depression. Am Psychol. 1973 Oct;28(10):857-70. doi: 10.1037/h0035605. No abstract available. PMID 4753644
- [Background] Fees BS, Martin P, Poon LW. A model of loneliness in older adults. J Gerontol B Psychol Sci Soc Sci. 1999 Jul;54(4):P231-9. doi: 10.1093/geronb/54b.4.p231. PMID 12382592
- [Background] Davidson EJ, Taylor CT, Ayers CR, Quach NE, Tu XM, Lee EE. The Relationship Between Loneliness and Positive Affect in Older Adults. Am J Geriatr Psychiatry. 2022 Jun;30(6):678-685. doi: 10.1016/j.jagp.2021.11.002. Epub 2021 Nov 12. PMID 34887211
- [Background] Compernolle EL, Finch LE, Hawkley LC, Cagney KA. Momentary loneliness among older adults: Contextual differences and their moderation by gender and race/ethnicity. Soc Sci Med. 2021 Sep;285:114307. doi: 10.1016/j.socscimed.2021.114307. Epub 2021 Aug 6. PMID 34375898
- [Background] Cohn MA, Pietrucha ME, Saslow LR, Hult JR, Moskowitz JT. An online positive affect skills intervention reduces depression in adults with type 2 diabetes. J Posit Psychol. 2014 Jan 1;9(6):523-534. doi: 10.1080/17439760.2014.920410. PMID 25214877
- [Background] Chou KL, Jun LW, Chi I. Assessing Chinese older adults' suicidal ideation: Chinese version of the Geriatric Suicide Ideation Scale. Aging Ment Health. 2005 Mar;9(2):167-71. doi: 10.1080/13607860412331336805. PMID 15804635
- [Background] Choi NG, Pepin R, Marti CN, Stevens CJ, Bruce ML. Improving Social Connectedness for Homebound Older Adults: Randomized Controlled Trial of Tele-Delivered Behavioral Activation Versus Tele-Delivered Friendly Visits. Am J Geriatr Psychiatry. 2020 Jul;28(7):698-708. doi: 10.1016/j.jagp.2020.02.008. Epub 2020 Mar 2. PMID 32238297
- [Background] Cheung EO, Cohn MA, Dunn LB, Melisko ME, Morgan S, Penedo FJ, Salsman JM, Shumay DM, Moskowitz JT. A randomized pilot trial of a positive affect skill intervention (lessons in linking affect and coping) for women with metastatic breast cancer. Psychooncology. 2017 Dec;26(12):2101-2108. doi: 10.1002/pon.4312. Epub 2016 Dec 27. PMID 27862646
- [Background] Chang Q, Sha F, Chan CH, Yip PSF. Validation of an abbreviated version of the Lubben Social Network Scale ("LSNS-6") and its associations with suicidality among older adults in China. PLoS One. 2018 Aug 2;13(8):e0201612. doi: 10.1371/journal.pone.0201612. eCollection 2018. PMID 30071067
- [Background] Cacioppo S, Grippo AJ, London S, Goossens L, Cacioppo JT. Loneliness: clinical import and interventions. Perspect Psychol Sci. 2015 Mar;10(2):238-49. doi: 10.1177/1745691615570616. PMID 25866548
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Barg FK, Huss-Ashmore R, Wittink MN, Murray GF, Bogner HR, Gallo JJ. A mixed-methods approach to understanding loneliness and depression in older adults. J Gerontol B Psychol Sci Soc Sci. 2006 Nov;61(6):S329-39. doi: 10.1093/geronb/61.6.s329. PMID 17114313
- [Background] Akhter-Khan SC, Prina M, Wong GH, Mayston R, Li L. Understanding and Addressing Older Adults' Loneliness: The Social Relationship Expectations Framework. Perspect Psychol Sci. 2023 Jul;18(4):762-777. doi: 10.1177/17456916221127218. Epub 2022 Nov 2. PMID 36322145